CLINICAL TRIAL: NCT06133894
Title: Effect of Exercise-education Program Inspired by Developmental Kinesiology on Determinants of Sarkopenia and Frailty in Late Life
Brief Title: Effect of Exercise-education Program PERMANENTO in Late Life
Acronym: PERMANENTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Vladimíra Dostálová, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NU22-09-00447
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Frailty; Sarcopenia
Keywords: prevention; older adults; functional status; frailty; sarcopenia; exercise; on-line program; sustainability
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of volunteers over 70 years of age
Who Masked: Outcomes Assessor
Masking Description: Single blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group was educated and instructed and agaged in a 12-week exercise program - 15 minutes 6 times per week of complex daily routines delivered via on-line platform.
  Interventions: Behavioral: Exercise program PERMANENTO inspired by developmental kinesiology
- Contol group (No Intervention): The control group continued in regular daily activities and was offered the same intervention as the experimental group after the research trial.

INTERVENTIONS:
Behavioral: Exercise program PERMANENTO inspired by developmental kinesiology — The intervention is based on activation of reflexive movement patterns which ensures the original reflexive control of strength, mobility and stability. After birth, we cannot control our body movements - they are reflexes "hard-wired" into our brains and vitally important for proper development of our body (muscular system, vestibular system, sensory system, cardiovascular system or digestive system) as well as our brain and nervous systems. During early childhood, everything becomes integrated and works perfectly according to the original design. But this design is slowly abandoned due to for example sedentary lifestyle and replaced by compensatory movement patterns that are making us weaker and defective with all the consequences that are becoming more severe as we age. The aim is restore the original design and improve posture and other crucial components of functional fitness and move better and more.
  Arms: Experimental group

SUMMARY:
The general aim of the present study is to create and empirically evaluate (RCT trial) an online education and exercise program (called PERMANENTO) to help older adults to understand the wider consequences of being active and offer them easy to follow exercise program inspired by developmental kinesiology.

DETAILED DESCRIPTION:
There is no doubt about the importance of a physical activity at a later age, yet it is often missing in the lives of seniors and the current epidemiological situation deepens this deficit even further. It is known that insufficient physical activity has a major effect on the decline of functional fitness components, premature development of sarcopenia or frailty syndrome, threatening self-sufficiency, health and consequently quality of life. This is associated with an increased burden on the health care system and related social services, with implications for public budgets. The aim of this project is to eliminate the onset or premature manifestation of negative aspects of aging by prevention. The content is to research a unique intervention inspired by the principles of developmental kinesiology with a presumed positive effect on the health status and the development of a comprehensive exercise and educational program for older adults. The main planned result of the project is a methodological manual and a web application containing education and exercise program for both older adults as well healthcare professionals.

The project responds to the priorities of the Applied Health Research Program for the years 2020-2026 and its focus contributes to a long-term solution of the population aging issue. With regard to demographic change, health and social care systems will be unsustainable without the adoption of preventive measures by seniors themselves. Exercise-educational intervention can lead to lasting changes and can help seniors to actively and responsibly participate in the course of their own aging. Main objective: to reduce negative health related aspects of aging, resp. their premature manifestation, by a preventive exercise-educational program. Sub-objectives: - to develop a specifically targeted exercise-educational program; - to demonstrate effectiveness of the program on health and social related indicators; - to assess acceptability, sustainability and other personal contexts - to create a methodological manual and a web platform for home-dwelling as well as institutionalized older adults containing complex information for independent exercise (how, as well as why).

ELIGIBILITY:
Inclusion Criteria:

* permanent residency in Prague
* being at least 70 years of age or older
* living independently at home

Exclusion Criteria:

* significant mobility limitation
* any health condition preventing from physical activity

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Timed up-and go test | Within a week prior the intervention and within a week after the intervention
  Performance-based measure of functional mobility and balance in older adults.The test requires the participant to rise from a chair, walk 3.0 m at a comfortable pace to a mark placed on the floor, turn around at the 3.0 m mark, walk back to the starting point, and return to sitting in the chair. The test's score is the time it takes the subject takes to complete the test. Lower score is better result.
Limits of stability on NeuroCom | Within a week prior the intervention and within a week after the intervention
  The Limits of Stability (LOS) test quantifies the maximum distance participant can lean own body (i.e. intentionally weight shift) in a given direction without losing balance, stepping, or reaching for assistance as would be required for function and gait. The scores for each parameter and movement direction are represented by a numeric value. Higher score is better result.
The Sensory Organization Test on NeuroCom | Within a week prior the intervention and within a week after the intervention
  The Sensory Organization Test (SOT) objectively identifies abnormalities in the patient's use of the three sensory systems that contribute to postural control: somatosensory, visual, and vestibular. The scores summarize the overall function of the three systems and the ability to resolve conflicting sensory inputs. Scores range from 0 to 100 (higher score, better result). Composite score identifies the presence of a balance control problem. Scores range from 0 to 100 (higher score, better result).
Body composition on InBody 720 | Within a week prior the intervention and within a week after the intervention
  The multifrequency body composition analyser InBody720 analyses body composition via the method of bioelectrical impedance (DSM-BIA) for every part of the body using 6 different frequencies (1kHz, 5kHz, 50kHz, 250kHz, 500kHz, 1000kHz) in each one of the five parts of the body with the quadrupole 8-point tactile system. It provides wide range of outcomes (main focus on: Body fat mass - lower score, better result, Skeletal muscle mass - higher score, better result, Visceral Fat - lower score, better result).
Handgrip strength on dynanometr | Within a week prior the intervention and within a week after the intervention
  Handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles. Participant is instructed to squeezes the dynamometer with maximum isometric effort, which is maintained for about 5 seconds. No other body movement is allowed. Higher score, better result.
Perceived functional fitness and health status | Within a week prior the intervention and within a week after the intervention
  Measured by questions "In general, would you say your health is poor, fair, good, very good, or excellent?" and "In general, would you say your functional fitness is poor, fair, good, very good, or excellent?". Score are represented on 5-point scale: (1) Excellent, 2) Very Good, 3) Good, 4) Fair, or 5) Poor). Lower score, better result.

SECONDARY OUTCOMES:
Long-term sustainability | 6 and 12 months after the end of the intervention
  To evaluate acceptance and long-term sustainability of the program via on-line questionnaire distributed among participants. The questionnaire is rather qualitative and includes Yes vs. No answers and open ended item.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Machacova, Principal Investigator — Centre of Expertise in Longevity and Long-term care, Faculty of Humanities, Charles University
Locations (1):
- Centre of Expertise oi Longevity and Long-term Care, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No